CLINICAL TRIAL: NCT05116540
Title: A Randomized, Double-Blind, Single-Center, Phase 2, Efficacy and Safety Study of Autologous HB-adMSCs vs Placebo for the Treatment of Patients With Multiple Sclerosis
Brief Title: Randomized Double-Blind Phase 2 Efficacy and Safety of Autologous HB-MSCs vs Placebo for Treatment of Multiple Sclerosis
Acronym: HBMS01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBMS01
Record Dates: First submitted 2021-10-27; First posted 2021-11-11 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Mesenchymal Stem Cells; MS; RRMS; stem cells; MSCs; Relapsing; Remitting
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded Randomized Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Adipose derived Mesenchymal stem cells (Autologous)
  Interventions: Biological: HB-adMSCs
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HB-adMSCs — Autologous product
  Other Names: Hope Biosciences adipose derived mesenchymal stem cells
  Arms: Treatment
Drug: Placebo — Normal Saline
  Other Names: 0.9% NS
  Arms: Placebo

SUMMARY:
Randomized Double-Blind Efficacy and safety study of Autologous HB-adMSCs versus placebo for the treatment of Multiple Sclerosis. This study will be for 24 subjects with 6 infusions over a 52 week period. Study participants will continue their established concomitant medications during participation in this investigation.

DETAILED DESCRIPTION:
Each eligible study subject will receive a total of 6 intravenous infusions of HB-adMSCs or placebo. Study infusions will be administered with the following regimen, Week 0, 4, 8, 16, 24, and 32. There will be one follow-up visit and end of study at week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18 - 75 years of age.
2. Study participants must have been diagnosed with Relapsing-Remitting Multiple Sclerosis (RRMS) for at least 6 months before study participation.
3. Study participants must be stabilized on any MS therapy for at least 6 months prior to randomization.
4. Study participants must agree not to increase or begin any Diseases Modifying Therapies for MS during participation in the clinical trial.
5. Study participants must have an EDSS score between 3.0 to 6.5. (Patient must be able to walk).
6. Study participants must have previously banked their mesenchymal stem cells with Hope Biosciences.
7. Study participants should be able to read, understand, and provide written consent.
8. Before any clinical-trial-related procedures are performed, informed consent must be obtained from the participants voluntarily.
9. Female study participants should not be pregnant or plan to become pregnant during study participation and for 6 months after last investigational product administration. *
10. Male participants, if their sexual partners can become pregnant, should use a method of contraception during study participation and for 6 months after the last administration of the investigated product. *
11. Study participant is able and willing to comply with the requirements of this clinical trial.
12. Participants in the study should have evidence of disease, as shown by MRIs of the brain or spinal cord, with the most recent being within 1 year of the screening date, and no other signs of relapse.

Exclusion Criteria:

1. Pregnancy, lactation. Women of childbearing age who are not pregnant but do not take effective contraceptive measures. *
2. Study participants with other types of multiple sclerosis, such as progressive relapsing, primary or secondary progressive.
3. Study participant has any active malignancy, including but not limited to evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
4. Study participant has known addiction or dependency or has current substance use or abuse.
5. Study participant has 1 or more significant concurrent medical conditions (verified by medical records), including the following:

   * Poorly controlled diabetes mellitus (PCDM) defined as history of deficient standard of care treatment and/or pre-prandial glucose >130mg/dl during screening visit or post-prandial glucose >200mg/dl.
   * Medical History of Chronic kidney disease (CKD) diagnosis and/or screening results of eGFR < 59mL/min/1.73m2.
   * Presence of New York Heart Association (NYHA) Class III/IV heart failure during screening visit.
   * Any medical history of myocardial infarction in any of the different types, such as ST-elevation myocardial infarction (STEMI) or non-ST-elevated myocardial infarction (NSTEMI), coronary spasm, or unstable angina.
   * Medical history of uncontrolled high blood pressure defined as a deficient standard of care treatment and/or blood pressure > 180/120 mm/Hg during screening visit.Medical history of diseases such as, inherited thrombophilias, cancer of the lung, brain, lymphatic, gynecologic system (ovary or uterus), or gastrointestinal tract (like pancreas or stomach).
   * Medical history of conditions, such as recent major general surgery, (within 12 months before the Screening), lower extremity paralysis due to spinal cord injury, fracture of the pelvis, hips, or femur.
6. Study participant has received any stem cell treatment within 12 months before first dose of investigational product other than stem cells produced by Hope Biosciences.
7. The study participant has received any experimental drug within 12 months before the first dose of the investigational product. (Except for COVID-19 vaccinations)
8. Study participant has a laboratory abnormality during screening, including the following:

   * White blood cell count < 3000/mm3
   * Platelet count < 80,000mm3
   * Absolute neutrophil count < 1500/mm3
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 10 upper limit of normal (ULN) x 1.5
9. Study participant has any other laboratory abnormality or medical condition which, in the opinion of the investigator poses a safety risk or will prevent the subject from completing the study.
10. The study participant has any concurrent neurologic disease, including hereditary conditions that the principal investigator considers could interfere with the study participation. Some of these neurologic diseases could be Charcot-Marie-Tooth (CMT) or Spinocerebellar Ataxia (SCA).
11. Study participant has any ongoing infection, including TB, CMV, EBV, HSV, VZV, hepatitis virus, toxoplasmosis, HIV, or syphilis infections, as well as hepatitis B surface antigen positive, and or/ hepatitis C PCR positivity.
12. Study participant is unlikely to complete the study or adhere to the study procedures.
13. Study participant has a previously diagnosed psychiatric condition which in the opinion of the investigator may affect self-assessments.
14. Study participants with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days prior to first dose of the investigational product.
15. Male study participants who plan to donate sperm during the study or within 6 months after the last dose. Female patients who plan to donate eggs or undergo in vitro fertilization treatment during the study or within 6 months after the last dose.
16. Study participants who are determined by the Investigator to be unsuitable for study enrollment for other reasons.
17. Participants' life expectancy must not have been considerably limited by other comorbidities, a history of previous myelodysplasia, or hematologic illness.

    * Acceptable reversible and permanent methods of birth control include:

1. True sexual abstinence (abstaining from sexual activity during the entire period of risk).

2. Surgery (occlusion bilateral tubal ligation, vasectomized partner). 3. Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable patch, or intravaginal). 4. Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data at this time

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Autologous Hope Biosciences adipose derived mesenchymal stem cells. HB-adMSCs: HB-adMSCs will be administered intravenously to study participants who qualify.
  Placebo: Placebo will be administered intravenously to study participants who qualify.
- Placebo: Sterile Saline Solution 0.9% HB-adMSCs: HB-adMSCs will be administered intravenously to study participants who qualify.
  Placebo: Placebo will be administered intravenously to study participants who qualify.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.57) | 49.1 (12.17) | 50.0 (11.19)
Age, Customized [Mean (Standard Deviation); unit: years] | 51.0 (10.57) | 49.1 (12.17) | 50.0 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Weight [Mean (Standard Deviation); unit: kilograms] | 68.61 (17.493) | 76.55 (16.619) | 72.58 (17.172)
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.72 (5.520) | 27.17 (5.723) | 25.94 (5.639)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Physical Health Composite Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  The developers used the SF-36 as a base and added 18 questions to address MS-specific problems, including fatigue and cognitive function.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function. There is no single overall score for MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
Time Frame: Baseline to Week 52
Population: One patient from the treatment group was unable to attend their follow-up visit (Week 42) and therefore was unable to complete the MSQOL-54 for that visit.
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 53.85 (9.61) | 44.07 (10.95)
  Infusion 3 (Week 8) | 8.21 (13.08) | 7.03 (10.76)
  Infusion 5 (Week 24) | 6.68 (7.33) | 3.43 (11.00)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 4.19 (18.03) | 0.06 (11.13)
  End of Study (Week 52) | 15.98 (12.08) | 2.03 (10.62)

2. Primary Outcome: Change From Baseline in Mental Health Composite Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 65.37 (24.83) | 60.88 (20.58)
  Infusion 3 (Week 8) | 11.04 (10.96) | 6.39 (21.55)
  Infusion 5 (Week 24) | 8.81 (11.20) | 3.22 (13.29)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 5.48 (17.96) | -0.35 (22.40)
  End of Study (Week 52) | 13.54 (15.65) | -2.59 (22.21)

3. Primary Outcome: Change From Baseline in Cognitive Function Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Cognitive Function subscale. The score ranges from 0 to 100 percent, and is 15% of the total Mental Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 59.55 (39.27) | 64.50 (36.32)
  Infusion 3 (Week 8) | 10.45 (23.29) | 6.50 (16.67)
  Infusion 5 (Week 24) | 5.91 (10.91) | 5.50 (14.80)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 3.00 (20.84) | 4.50 (17.55)
  End of Study (Week 52) | 9.55 (18.09) | -2.50 (10.07)

4. Primary Outcome: Change From Baseline in Emotional Well-Being Composite Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Emotional Wellbeing sub-scale. The score ranges from 0 to 100 percent, and is 29% of the total Mental Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 71.27 (21.45) | 68.40 (17.23)
  Infusion 3 (Week 8) | 6.91 (14.32) | 3.60 (11.54)
  Infusion 5 (Week 24) | 6.55 (10.47) | 3.20 (13.31)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 4.80 (21.81) | 2.40 (12.82)
  End of Study (Week 52) | 12.36 (17.66) | -1.20 (11.63)

5. Primary Outcome: Change From Baseline in Health Distress Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Health Distress sub-scale. The score ranges from 0 to 100 percent, and is 14% of the total Mental Health Composite Score and 11% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 54.09 (24.58) | 36.00 (28.07)
  Infusion 3 (Week 8) | 19.55 (25.44) | 16.50 (22.12)
  Infusion 5 (Week 24) | 13.18 (25.33) | 4.50 (19.36)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 5.50 (40.03) | 2.50 (19.18)
  End of Study (Week 52) | 25.00 (28.55) | -2.00 (13.58)

6. Primary Outcome: Change From Baseline in RL/Emotional Problems Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Role Limitation/Emotional sub-scale. The score ranges from 0 to 100 percent, and is 24% of the total Mental Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 63.64 (43.35) | 73.33 (43.89)
  Infusion 3 (Week 8) | 15.15 (27.34) | 3.33 (65.64)
  Infusion 5 (Week 24) | 15.15 (27.34) | 0.00 (41.57)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 13.33 (28.11) | -10.00 (66.76)
  End of Study (Week 52) | 18.18 (31.14) | -10.00 (80.20)

7. Primary Outcome: Change From Baseline in Overall Quality of Life Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Overall Quality of Life sub-scale. The score ranges from 0 to 100 percent, and is 18% of the total Mental Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 71.82 (15.92) | 48.50 (12.62)
  Infusion 3 (Week 8) | 6.05 (13.93) | 7.00 (12.55)
  Infusion 5 (Week 24) | 3.04 (14.20) | 4.67 (12.15)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | -1.83 (14.54) | 1.84 (12.52)
  End of Study (Week 52) | 3.64 (10.14) | 4.50 (9.85)

8. Primary Outcome: Change From Baseline in Energy/Fatigue Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Energy/Fatigue sub-scale. The score ranges from 0 to 100 percent, and is 12% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 48.00 (15.59) | 32.00 (21.08)
  Infusion 3 (Week 8) | 6.18 (13.67) | 13.60 (14.14)
  Infusion 5 (Week 24) | 4.36 (17.75) | 10.40 (14.01)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 2.00 (21.44) | 2.40 (17.40)
  End of Study (Week 52) | 15.27 (20.62) | 1.60 (9.47)

9. Primary Outcome: Change From Baseline in Health Perception Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Health Perception sub-scale. The score ranges from 0 to 100 percent, and is 17% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 59.55 (18.09) | 42.00 (21.76)
  Infusion 3 (Week 8) | 9.09 (18.68) | 5.00 (9.43)
  Infusion 5 (Week 24) | 0.00 (17.03) | 3.50 (15.82)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 10.00 (15.09) | -1.50 (12.48)
  End of Study (Week 52) | 12.27 (19.41) | -2.00 (12.06)

10. Primary Outcome: Change From Baseline in Physical Function Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Physical Function sub-scale. The score ranges from 0 to 100 percent, and is 17% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 36.36 (25.21) | 43.00 (17.19)
  Infusion 3 (Week 8) | 1.36 (24.20) | -1.50 (15.28)
  Infusion 5 (Week 24) | 12.27 (10.09) | -6.00 (19.26)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 7.50 (13.99) | -0.50 (19.78)
  End of Study (Week 52) | 7.73 (15.06) | 7.00 (25.63)

11. Primary Outcome: Change From Baseline in RL/Physical Problems Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Role Limitations - Physical sub-scale. The score ranges from 0 to 100 percent, and is 12% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 38.64 (40.87) | 20.00 (32.91)
  Infusion 3 (Week 8) | 11.36 (42.37) | 22.50 (38.10)
  Infusion 5 (Week 24) | 6.82 (38.88) | 17.50 (35.45)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | -2.50 (49.23) | 5.00 (15.81)
  End of Study (Week 52) | 34.09 (45.10) | 10.00 (50.28)

12. Primary Outcome: Change From Baseline in Pain Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Pain subscale. The score ranges from 0 to 100 percent, and is 11% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 71.82 (14.38) | 59.83 (27.66)
  Infusion 3 (Week 8) | 7.12 (15.19) | 7.17 (17.02)
  Infusion 5 (Week 24) | 4.55 (26.28) | 4.34 (16.80)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | -1.50 (32.12) | 0.00 (14.66)
  End of Study (Week 52) | 13.49 (18.17) | 1.33 (17.65)

13. Primary Outcome: Change From Baseline in Social Function Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Social Function subscale. The score ranges from 0 to 100 percent, and is 12% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 67.42 (23.70) | 59.17 (14.93)
  Infusion 3 (Week 8) | 6.06 (25.02) | -2.50 (11.15)
  Infusion 5 (Week 24) | 5.30 (13.58) | -1.67 (15.11)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 2.50 (23.26) | -4.16 (27.00)
  End of Study (Week 52) | 13.64 (25.35) | 1.67 (15.11)

14. Primary Outcome: Change From Baseline in Sexual Function Score - Multiple Sclerosis Quality of Life (MSQOL) 54 Instrument.
Description: The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function, and each one is scored from 0 to 100. Two summary scores - physical health and mental health - can be derived from a weighted summation of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).
  This outcome measure shows the change from baseline of the Sexual Function subscale. The score ranges from 0 to 100 percent, and is 8% of the total Physical Health Composite Score.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total)
  Infusion 1/Baseline (Week 0) | 65.15 (30.47) | 71.67 (24.60)
  Infusion 3 (Week 8) | 8.33 (25.27) | -2.50 (20.44)
  Infusion 5 (Week 24) | 8.34 (26.09) | -3.33 (20.87)
  Follow-Up (Week 42): number analyzed (Participants) | 10 | 10
  Follow-Up (Week 42) | 6.66 (33.52) | -3.33 (14.28)
  End of Study (Week 52) | 9.85 (19.65) | -4.16 (15.84)

15. Primary Outcome: Analysis of Covariance (ANCOVA) Model - Physical Health Composite Score Change From Baseline Multiple Sclerosis Quality of Life (MSQOL)-54
Description: Analysis of covariance (ANCOVA) is a statistical model that combines linear regression and ANOVA to analyze the results of different treatments. In this outcome measure, ANCOVA was used to analyze change in the physical health composite score in treatment versus placebo. The ANCOVA model was used to compare HB-adMSC patients with placebo patients on Change from Baseline to Week 52 with a fixed factor of treatment, fixed stratification factors of MS severity, age and gender, and a covariate of the baseline value for the score on the corresponding outcome measure. This model allows us to test the significance of the effects of the treatment at Week 52. Total score for this subscale is 100, so the range of scores for the ANCOVA model (showing average change in scores) would be -100 to 100 (theoretically). Higher scores show better outcomes--in this model, a positive score would indicate improvement and a negative score indicates worsening. Subscales are interpreted separately.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total) | 19.872 (2.979) | -2.248 (3.145)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 22.121, 95% CI 2-sided [12.282 to 31.959], Standard Error of Mean 4.616

16. Primary Outcome: Analysis of Covariance (ANCOVA) Model - Mental Health Composite Score Change From Baseline Multiple Sclerosis Quality of Life (MSQOL)-54 Composite Score
Description: Analysis of covariance (ANCOVA) is a statistical model that combines linear regression and ANOVA to analyze the results of different treatments. In this outcome measure, ANCOVA was used to analyze change in the mental health composite score in treatment versus placebo. The ANCOVA model was used to compare HB-adMSC patients with placebo patients on Change from Baseline to Week 52 with a fixed factor of treatment, fixed stratification factors of MS severity, age and gender, and a covariate of the baseline value for the score on the corresponding outcome measure. This model allows us to test the significance of the effects of the treatment at Week 52. Total score for this subscale is 100, so the range of scores for the ANCOVA model (showing average change in scores) would be -100 to 100 (theoretically). Higher scores show better outcomes--in this model, a positive score would indicate improvement and a negative score indicates worsening. Subscales are interpreted separately.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total) | 13.362 (3.961) | -2.402 (4.161)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0166, ANCOVA; Mean Difference (Final Values) = 15.764, 95% CI 2-sided [3.307 to 28.221], Standard Error of Mean 5.844

17. Primary Outcome: Bayesian Statistical Analysis - Analysis of Covariance (ANCOVA) Model - Physical Health Composite Score Change From Baseline Multiple Sclerosis Quality of Life (MSQOL)-54
Description: Bayesian analysis is a statistical method that uses probability distributions to make statistical inferences about parameters using prior information. In this outcome measure, Bayesian analysis was used to analyze change in the physical health composite score in treatment versus placebo. In this study, Bayesian analysis was used to estimate the posterior distribution and to estimate the probability of the true treatment difference of change from baseline to Week 52. A linear model for each visit was constructed to model within-subject observation covariance structures by multivariate normal (MVN) distribution in the Markov chain Monte Carlo (MCMC) procedure. Total score for this subscale is 100, so the range of scores for the ANCOVA model (showing average change in scores) would be -100 to 100 (theoretically). Higher scores show better outcomes--in this model, a positive score would indicate improvement and a negative score indicates worsening. Subscales are interpreted separately.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total) | 18.373 (5.426) | -3.764 (5.308)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.9905, ANCOVA; Mean Difference (Final Values) = 22.137, 95% CI 2-sided [12.361 to 32.006], Standard Deviation 4.962

18. Primary Outcome: Bayesian Statistical Analysis - Analysis of Covariance (ANCOVA) Model - Mental Health Composite Score Change From Baseline - Multiple Sclerosis Quality of Life (MSQOL)-54
Description: Bayesian analysis is a statistical method that uses probability distributions to make statistical inferences about parameters using prior information. In this outcome measure, Bayesian analysis was used to analyze change in the mental health composite score in treatment versus placebo. In this study, Bayesian analysis was used to estimate the posterior distribution and to estimate the probability of the true treatment difference of change from baseline to Week 52. A linear model for each visit was constructed to model within-subject observation covariance structures by multivariate normal (MVN) distribution in the Markov chain Monte Carlo (MCMC) procedure. Total score for this subscale is 100, so the range of scores for the ANCOVA model (showing average change in scores) would be -100 to 100 (theoretically). Higher scores show better outcomes--in this model, a positive score would indicate improvement and a negative score indicates worsening. Subscales are interpreted separately.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (100 points total) | 12.414 (7.457) | -3.333 (7.544)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.8292, ANCOVA; Mean Difference (Final Values) = 15.747, 95% CI 2-sided [3.329 to 28.177], Standard Deviation 6.274

19. Secondary Outcome: Analysis of Covariance (ANCOVA) Model - Total Expanded Disability Status Scale (EDSS) Scores Through Week 52 - Change From Baseline - Efficacy Analysis Set
Description: The EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. This scale ranges from 0 to 10 in 0.5-unit increments and a higher score represents increased disability. Scoring is based on an examination by a neurologist.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Groups:
- Treatment: Autologous Hope Biosciences adipose derived mesenchymal stem cells. HB-adMSCs: HB-adMSCs will be administered intravenously to study participants who qualify.
- Placebo: Sterile Saline Solution 0.9%
  Placebo: Placebo will be administered intravenously to study participants who qualify.
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (10 points total) | -1.502 (0.424) | 0.052 (0.446)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0278, ANCOVA; Mean Difference (Final Values) = -1.554, 95% CI 2-sided [-2.914 to -0.195], Standard Error of Mean 0.638

20. Secondary Outcome: Analysis of Covariance (ANCOVA) Model - Change From Baseline Barthel Index Scores Through Week 52 - Efficacy Analysis Set
Description: The Barthel index is an ordinal scale that evaluates functional independence in the domains of personal care and mobility. A total of ten variables describing activities of daily living and mobility are considered, with a higher number reflecting better capacity to operate independently. The Barthel Index assesses the level of help needed by a person on a set of ten activities of daily living (ADL) related to mobility and self-care. Score ranges from 0 points to 20 points, with lower scores indicating increased disability.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: score on a scale (20 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (20 points total) | 2.359 (1.867) | -3.094 (1.962)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0666, ANCOVA; Mean Difference (Final Values) = 5.453, 95% CI 2-sided [-0.424 to 11.330], Standard Error of Mean 2.757

21. Secondary Outcome: ANCOVA Model - Change From Baseline 9-Hole Peg Test Scores - Dominant Hand Avg Time Through Week 52
Description: The 9-HPT is a short, standardized upper extremity exam. It measures the time taken to complete the test activity, recorded in seconds. The higher the score the worse the disability.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
seconds | 0.472 (3.725) | -9.639 (3.915)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0863, ANCOVA; Mean Difference (Final Values) = 10.112, 95% CI 2-sided [-1.629 to 21.853], Standard Error of Mean 5.508

22. Secondary Outcome: Analysis of Covariance (ANCOVA) Model - Change From Baseline 9-Hole Peg Test Scores - Non-Dominant Hand Avg Time Through Week 52
Description: as for outcome 21
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
seconds | -3.771 (1.069) | -4.747 (1.127)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.5588, ANCOVA; Mean Difference (Final Values) = 0.977, 95% CI 2-sided [-2.504 to 4.457], Standard Error of Mean 1.633

23. Secondary Outcome: Analysis of Covariance (ANCOVA) Model - Change in Patient Health Questionnaire (PHQ-9) Test Scores
Description: The PHQ-9 is the most used depression and suicidal thoughts screening test used to monitor the severity of depression and response to treatment. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Error); unit: score on a scale (27 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale (27 points total) | -4.330 (0.693) | 0.263 (0.728)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -4.593, 95% CI 2-sided [-6.773 to -2.413], Standard Error of Mean 1.023

24. Secondary Outcome: Baseline Vitals Values - Height
Description: Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline
Measure: Mean (Standard Error); unit: cm
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
cm | 166.17 (3.151) | 167.86 (2.626)

25. Secondary Outcome: Change From Baseline Vitals Values - Weight
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: One patient from the treatment group was unable to attend starting at their follow-up visit (Week 42), and two patients from the Placebo group stopped attending visits starting at their Infusion 5 visit (Week 24) .
Measure: Mean (Standard Error); unit: kg
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
kg
  Infusion 1 (Baseline) | 68.61 (5.050) | 76.55 (4.797)
  Infusion 2 - Week 4 | 0.15 (0.309) | 0.18 (0.406)
  Infusion 3- Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3- Week 8 | -0.04 (0.385) | -0.05 (0.441)
  Infusion 4- Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4- Week 16 | 1.02 (0.972) | -0.18 (0.727)
  Infusion 5- Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5- Week 24 | 0.56 (1.043) | -0.56 (0.923)
  Infusion 6- Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6- Week 32 | 1.05 (1.105) | -0.31 (1.149)
  Follow-Up- Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up- Week 42 | 1.19 (2.665) | -0.14 (1.350)
  End of Study- Week 52: number analyzed (Participants) | 11 | 10
  End of Study- Week 52 | 0.82 (1.519) | 0.03 (1.332)

26. Secondary Outcome: Change From Baseline Vitals Values - Body Mass Index
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2
  Infusion 1 (Baseline) | 24.72 (1.593) | 27.17 (1.652)
  Infusion 2 - Week 4 | 0.05 (0.112) | 0.07 (0.146)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | -0.00 (0.142) | -0.04 (0.164)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | 0.46 (0.399) | -0.05 (0.263)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | 0.28 (0.417) | -0.19 (0.332)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | 0.47 (0.436) | -0.11 (0.399)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | 0.61 (1.014) | -0.05 (0.476)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | 0.37 (0.591) | -0.02 (0.505)

27. Secondary Outcome: Change From Baseline Vitals Values - Respiratory Rate
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: Breaths/min
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Breaths/min
  Infusion 1 (Baseline) | 16.7 (0.28) | 16.3 (0.22)
  Infusion 2 - Week 4 | 0.0 (0.35) | 0.2 (0.17)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | 0.0 (0.35) | 0.4 (0.24)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | 0.0 (0.00) | 0.5 (0.28)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | -0.2 (0.17) | 0.6 (0.31)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | 0.2 (0.17) | 0.2 (0.20)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | 0.4 (0.24) | 0.6 (0.31)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | 0.2 (0.33) | 0.6 (0.31)

28. Secondary Outcome: Change From Baseline Vitals Values - Temperature
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: degrees Celsius
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
degrees Celsius
  Infusion 1 (Baseline) | 36.66 (0.073) | 36.84 (0.080)
  Infusion 2 - Week 4 | -0.01 (0.083) | -0.23 (0.070)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | 0.03 (0.095) | -0.21 (0.108)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | -0.03 (0.074) | -0.06 (0.095)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | 0.04 (0.084) | -0.17 (0.115)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | -0.08 (0.102) | -0.18 (0.101)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | -0.10 (0.077) | -0.15 (0.092)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | -0.02 (0.088) | -0.11 (0.132)

29. Secondary Outcome: Change From Baseline Vitals Values - Systolic Blood Pressure
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
mmHg
  Infusion 1 (Baseline) | 119.2 (2.90) | 122.2 (3.72)
  Infusion 2 - Week 4 | 6.3 (3.10) | 0.8 (2.74)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | -5.0 (2.11) | -2.8 (3.62)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | 1.5 (3.27) | 5.4 (3.25)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | -3.5 (3.18) | -0.6 (2.77)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | 4.3 (3.87) | 1.5 (3.37)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | -4.0 (3.83) | -1.1 (2.52)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | 1.4 (4.43) | 0.7 (4.26)

30. Secondary Outcome: Change From Baseline Vitals Values - Diastolic Blood Pressure
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
mmHg
  Infusion 1 (Baseline) | 76.3 (1.90) | 78.9 (1.53)
  Infusion 2 - Week 4 | 2.5 (2.00) | 1.1 (1.91)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | -1.3 (1.97) | 0.0 (2.23)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | 0.9 (2.66) | 2.4 (2.21)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | -3.2 (2.17) | 1.4 (1.97)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | 4.0 (1.85) | 2.6 (2.93)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | -1.6 (2.76) | 3.6 (3.11)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | -1.1 (2.27) | 3.3 (2.12)

31. Secondary Outcome: Change From Baseline Vitals Values - Pulse Rate
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
beats per minute
  Infusion 1 (Baseline) | 71.8 (3.16) | 76.2 (1.66)
  Infusion 2 - Week 4 | 0.4 (2.60) | -0.9 (2.00)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | 3.3 (3.40) | 2.4 (2.57)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | 0.3 (3.70) | 2.0 (2.38)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | -2.6 (2.71) | -1.1 (2.22)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | 1.9 (4.30) | -2.1 (2.25)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 12
  Follow-Up - Week 42 | 1.2 (3.30) | -4.0 (2.56)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | -4.1 (2.48) | -1.2 (3.21)

32. Secondary Outcome: Change From Baseline Vitals Values - Oxygen Saturation
Description: Change From Baseline Vitals by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: as for outcome 25
Measure: Mean (Standard Error); unit: percent of oxygen
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
percent of oxygen
  Infusion 1 (Baseline) | 98.4 (0.23) | 98.0 (0.35)
  Infusion 2 - Week 4 | -0.7 (0.40) | 0.6 (0.38)
  Infusion 3 - Week 8: number analyzed (Participants) | 12 | 11
  Infusion 3 - Week 8 | -0.4 (0.38) | 0.5 (0.45)
  Infusion 4 - Week 16: number analyzed (Participants) | 12 | 11
  Infusion 4 - Week 16 | -0.4 (0.34) | 0.3 (0.47)
  Infusion 5 - Week 24: number analyzed (Participants) | 12 | 10
  Infusion 5 - Week 24 | 0.0 (0.30) | -0.4 (0.31)
  Infusion 6 - Week 32: number analyzed (Participants) | 12 | 10
  Infusion 6 - Week 32 | -0.9 (0.54) | 0.3 (0.47)
  Follow-Up - Week 42: number analyzed (Participants) | 11 | 10
  Follow-Up - Week 42 | -0.4 (0.28) | -0.5 (0.64)
  End of Study - Week 52: number analyzed (Participants) | 11 | 10
  End of Study - Week 52 | -0.5 (0.45) | 0.4 (0.54)

33. Secondary Outcome: Change From Baseline Physical Examination Results - Abdomen
Description: Change From Baseline Physical Examination Results by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 12 | 12
  Infusion 1 (Baseline): Abnormal | 0 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 12 | 11
  Infusion 3 - Week 8: Abnormal | 0 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 10
  Follow-Up - Week 42: Abnormal | 0 | 0
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

34. Secondary Outcome: Change From Baseline Physical Examination Results - Cardiovascular
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 12 | 12
  Infusion 1 (Baseline): Abnormal | 0 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 12 | 11
  Infusion 3 - Week 8: Abnormal | 0 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 10
  Follow-Up - Week 42: Abnormal | 0 | 0
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

35. Secondary Outcome: Change From Baseline Physical Examination Results - HEENT
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 12 | 12
  Infusion 1 (Baseline): Abnormal | 0 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 12 | 11
  Infusion 3 - Week 8: Abnormal | 0 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 10
  Follow-Up - Week 42: Abnormal | 0 | 0
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

36. Secondary Outcome: Change From Baseline Physical Examination Results - Lymph Node
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 12 | 12
  Infusion 1 (Baseline): Abnormal | 0 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 12 | 11
  Infusion 3 - Week 8: Abnormal | 0 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 10
  Follow-Up - Week 42: Abnormal | 0 | 0
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

37. Secondary Outcome: Change From Baseline Physical Examination Results - Musculoskeletal
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 6 | 3
  Infusion 1 (Baseline): Abnormal | 6 | 9
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 7 | 4
  Infusion 2 - Week 4: Abnormal | 5 | 8
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 5 | 3
  Infusion 3 - Week 8: Abnormal | 7 | 8
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 5 | 4
  Infusion 4 - Week 16: Abnormal | 7 | 7
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 4 | 4
  Infusion 5 - Week 24: Abnormal | 8 | 6
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 4 | 4
  Infusion 6 - Week 32: Abnormal | 8 | 6
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 2 | 4
  Follow-Up - Week 42: Abnormal | 9 | 6
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 3 | 4
  End of Study - Week 52: Abnormal | 8 | 6
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

38. Secondary Outcome: Change From Baseline Physical Examination Results - Neurological
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 2 | 1
  Infusion 1 (Baseline): Abnormal | 10 | 11
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 3 | 1
  Infusion 2 - Week 4: Abnormal | 9 | 11
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 1 | 1
  Infusion 3 - Week 8: Abnormal | 11 | 10
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 1 | 1
  Infusion 4 - Week 16: Abnormal | 11 | 10
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 1 | 1
  Infusion 5 - Week 24: Abnormal | 11 | 9
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 2 | 2
  Infusion 6 - Week 32: Abnormal | 10 | 8
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 0 | 1
  Follow-Up - Week 42: Abnormal | 11 | 9
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 2 | 2
  End of Study - Week 52: Abnormal | 9 | 8
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

39. Secondary Outcome: Change From Baseline Physical Examination Results - Respiratory
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 12 | 12
  Infusion 1 (Baseline): Abnormal | 0 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 12 | 11
  Infusion 3 - Week 8: Abnormal | 0 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 10
  Follow-Up - Week 42: Abnormal | 0 | 0
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

40. Secondary Outcome: Change From Baseline Physical Examination Results - Skin
Description: Change From Baseline Physical Examination by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Infusion 1 (Baseline): Normal | 11 | 12
  Infusion 1 (Baseline): Abnormal | 1 | 0
  Infusion 1 (Baseline): Not Examined (No longer in Study) | 0 | 0
  Infusion 2 - Week 4: Normal | 12 | 12
  Infusion 2 - Week 4: Abnormal | 0 | 0
  Infusion 2 - Week 4: Not Examined (No longer in Study) | 0 | 0
  Infusion 3 - Week 8: Normal | 11 | 11
  Infusion 3 - Week 8: Abnormal | 1 | 0
  Infusion 3 - Week 8: Not Examined (No longer in Study) | 0 | 1
  Infusion 4 - Week 16: Normal | 12 | 11
  Infusion 4 - Week 16: Abnormal | 0 | 0
  Infusion 4 - Week 16: Not Examined (No longer in Study) | 0 | 1
  Infusion 5 - Week 24: Normal | 12 | 10
  Infusion 5 - Week 24: Abnormal | 0 | 0
  Infusion 5 - Week 24: Not Examined (No longer in Study) | 0 | 2
  Infusion 6 - Week 32: Normal | 12 | 10
  Infusion 6 - Week 32: Abnormal | 0 | 0
  Infusion 6 - Week 32: Not Examined (No longer in Study) | 0 | 2
  Follow-Up - Week 42: Normal | 11 | 9
  Follow-Up - Week 42: Abnormal | 0 | 1
  Follow-Up - Week 42: Not Examined (No longer in Study) | 1 | 2
  End of Study - Week 52: Normal | 11 | 10
  End of Study - Week 52: Abnormal | 0 | 0
  End of Study - Week 52: Not Examined (No longer in Study) | 1 | 2

41. Secondary Outcome: Laboratory Values - CBC (x10^3 Cells/uL)
Description: Unit (x10^3 cells/uL) - Change From Baseline Clinical Laboratory Complete Blood Count (CBC) by Treatment Week - Descriptive Statistics - Safety Analysis Set
Time Frame: Baseline to Week 52
Population: One patient from the treatment group was unable to attend their end of study visit (Week 52), and two patients from the Placebo group stopped attending visits from before their Infusion 5 visit (Week 24) .
Measure: Mean (Standard Error); unit: (x10^3 cells/uL)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
(x10^3 cells/uL)
  Absolute Basophils - Baseline | 0.027 (0.0048) | 0.030 (0.0051)
  Absolute Basophils - Week 24: number analyzed (Participants) | 12 | 10
  Absolute Basophils - Week 24 | 0.008 (0.0063) | 0.003 (0.0050)
  Absolute Basophils - Week 52: number analyzed (Participants) | 11 | 10
  Absolute Basophils - Week 52 | 0.008 (0.0064) | -0.001 (0.0053)
  Absolute Eosinophils - Baseline | 0.107 (0.0267) | 0.113 (0.0221)
  Absolute Eosinophils - Week 24: number analyzed (Participants) | 12 | 10
  Absolute Eosinophils - Week 24 | -0.001 (0.0172) | 0.018 (0.0156)
  Absolute Eosinophils - Week 52: number analyzed (Participants) | 11 | 10
  Absolute Eosinophils - Week 52 | 0.027 (0.0302) | 0.012 (0.0150)
  Absolute Lymphocytes - Baseline | 1.345 (0.0956) | 1.220 (0.1370)
  Absolute Lymphocytes - Week 24: number analyzed (Participants) | 12 | 10
  Absolute Lymphocytes - Week 24 | 0.098 (0.1275) | 0.061 (0.0631)
  Absolute Lymphocytes - Week 52: number analyzed (Participants) | 11 | 10
  Absolute Lymphocytes - Week 52 | 0.155 (0.1179) | 0.072 (0.0797)
  Absolute Monocytes - Baseline | 0.501 (0.0536) | 0.494 (0.0549)
  Absolute Monocytes - Week 24: number analyzed (Participants) | 12 | 10
  Absolute Monocytes - Week 24 | -0.030 (0.0479) | -0.008 (0.0296)
  Absolute Monocytes - Week 52: number analyzed (Participants) | 11 | 10
  Absolute Monocytes - Week 52 | 0.069 (0.0543) | 0.009 (0.0307)
  Absolute Neutrophils - Baseline | 3.348 (0.4070) | 3.872 (0.4055)
  Absolute Neutrophils - Week 24: number analyzed (Participants) | 12 | 10
  Absolute Neutrophils - Week 24 | 0.470 (0.4303) | -0.066 (0.5305)
  Absolute Neutrophils - Week 52: number analyzed (Participants) | 11 | 10
  Absolute Neutrophils - Week 52 | 0.681 (0.5759) | 0.201 (0.5813)
  Platelet Count - Baseline | 260.6 (20.61) | 227.1 (20.28)
  Platelet Count - Week 24: number analyzed (Participants) | 12 | 10
  Platelet Count - Week 24 | 1.1 (8.64) | 11.1 (11.83)
  Platelet Count - Week 52: number analyzed (Participants) | 11 | 10
  Platelet Count - Week 52 | 19.9 (8.45) | 9.5 (7.81)
  WBC - Baseline | 5.35 (0.447) | 5.75 (0.504)
  WBC - Week 24: number analyzed (Participants) | 12 | 10
  WBC - Week 24 | 0.54 (0.450) | 0.01 (0.512)
  WBC - Week 52: number analyzed (Participants) | 11 | 10
  WBC - Week 52 | 0.95 (0.577) | 0.30 (0.537)

42. Secondary Outcome: Laboratory Values - CBC (% of WBC)
Description: Changes from baseline in CBC laboratory values with unit of % of white blood cell count.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: % of white blood cell count
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
% of white blood cell count
  Basophils - Baseline | 0.40 (0.161) | 0.74 (0.192)
  Basophils - Week 24: number analyzed (Participants) | 12 | 10
  Basophils - Week 24 | 0.22 (0.292) | 0.09 (0.308)
  Basophils - Week 52: number analyzed (Participants) | 11 | 10
  Basophils - Week 52 | 0.03 (0.259) | -0.13 (0.256)
  Eosinophils - Baseline | 1.86 (0.552) | 2.02 (0.409)
  Eosinophils - Week 24: number analyzed (Participants) | 12 | 10
  Eosinophils - Week 24 | 0.18 (0.656) | 1.06 (0.861)
  Eosinophils - Week 52: number analyzed (Participants) | 11 | 10
  Eosinophils - Week 52 | -0.01 (0.591) | 0.42 (0.373)
  Lymphocytes - Baseline | 27.98 (3.068) | 24.41 (2.049)
  Lymphocytes - Week 24: number analyzed (Participants) | 12 | 10
  Lymphocytes - Week 24 | 1.58 (2.945) | 1.21 (3.152)
  Lymphocytes - Week 52: number analyzed (Participants) | 11 | 10
  Lymphocytes - Week 52 | -3.46 (2.907) | 1.77 (4.329)
  Monocytes - Baseline | 8.59 (1.046) | 9.10 (1.215)
  Monocytes - Week 24: number analyzed (Participants) | 12 | 10
  Monocytes - Week 24 | -0.15 (1.124) | -0.76 (1.735)
  Monocytes - Week 52: number analyzed (Participants) | 11 | 10
  Monocytes - Week 52 | 1.83 (1.166) | -0.02 (1.564)
  Neutrophils - Baseline | 61.17 (2.777) | 63.73 (2.516)
  Neutrophils - Week 24: number analyzed (Participants) | 12 | 10
  Neutrophils - Week 24 | -2.06 (3.201) | -1.68 (4.138)
  Neutrophils - Week 52: number analyzed (Participants) | 11 | 10
  Neutrophils - Week 52 | 1.38 (3.861) | -2.21 (5.063)

43. Secondary Outcome: Laboratory Values - CBC (% of Total Blood Cell Count)
Description: Changes from baseline in CBC laboratory values with unit of % of total blood cell count.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: % of total blood cell count
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
% of total blood cell count
  Hematocrit - Baseline | 39.80 (0.736) | 40.77 (1.111)
  Hematocrit - Week 24: number analyzed (Participants) | 12 | 10
  Hematocrit - Week 24 | -0.48 (1.064) | 1.43 (1.392)
  Hematocrit- Week 52: number analyzed (Participants) | 11 | 10
  Hematocrit- Week 52 | 1.02 (0.562) | 2.51 (1.116)

44. Secondary Outcome: Laboratory Values - CBC (g/dL)
Description: Changes from baseline in CBC laboratory values with unit of g/dL
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
g/dL
  Hemoglobin - Baseline | 13.60 (0.301) | 13.68 (0.410)
  Hemoglobin - Week 24: number analyzed (Participants) | 12 | 10
  Hemoglobin - Week 24 | -0.18 (0.281) | 0.61 (0.498)
  Hemoglobin- Week 52: number analyzed (Participants) | 11 | 10
  Hemoglobin- Week 52 | 0.21 (0.168) | 0.81 (0.401)
  MCHC - Baseline | 34.13 (0.233) | 33.53 (0.233)
  MCHC - Week 24: number analyzed (Participants) | 12 | 10
  MCHC - Week 24 | -0.01 (0.340) | 0.31 (0.312)
  MCHC- Week 52: number analyzed (Participants) | 11 | 10
  MCHC- Week 52 | -0.31 (0.236) | -0.06 (0.352)

45. Secondary Outcome: Laboratory Values - CBC (pg)
Description: Changes from baseline in CBC laboratory values with unit of pg
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: pg
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
pg
  MCH - Baseline | 31.20 (0.542) | 30.38 (0.471)
  MCH - Week 24: number analyzed (Participants) | 12 | 10
  MCH - Week 24 | -0.23 (0.371) | 0.50 (0.286)
  MCH- Week 52: number analyzed (Participants) | 11 | 10
  MCH- Week 52 | -0.25 (0.276) | 0.44 (0.465)

46. Secondary Outcome: Laboratory Values - CBC (fL)
Description: Changes from baseline in CBC laboratory values with unit of fL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: fL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
fL
  MCV - Baseline | 91.36 (1.332) | 90.59 (1.163)
  MCV - Week 24: number analyzed (Participants) | 12 | 10
  MCV - Week 24 | -0.60 (0.937) | 0.65 (0.447)
  MCV - Week 52: number analyzed (Participants) | 11 | 10
  MCV - Week 52 | 0.15 (0.900) | 1.32 (0.857)

47. Secondary Outcome: Laboratory Values - CBC (x10^6 Cells/uL)
Description: Changes from baseline in CBC laboratory values with unit of x10^6 cells/uL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: x10^6 cells/uL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
x10^6 cells/uL
  RBC - Baseline | 4.362 (0.0772) | 4.507 (0.1293)
  RBC - Week 24: number analyzed (Participants) | 12 | 10
  RBC - Week 24 | -0.027 (0.1130) | 0.134 (0.1769)
  RBC - Week 52: number analyzed (Participants) | 11 | 10
  RBC - Week 52 | 0.100 (0.0645) | 0.222 (0.1571)

48. Secondary Outcome: Laboratory Values - CBC (RDW)
Description: Changes from baseline in CBC laboratory values with unit of % (RDW - Red Cell Distribution Width)
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
percentage
  RDW - Baseline | 12.51 (0.337) | 12.82 (0.162)
  RDW - Week 24: number analyzed (Participants) | 12 | 10
  RDW - Week 24 | 0.21 (0.155) | 0.57 (0.585)
  RDW - Week 52: number analyzed (Participants) | 11 | 10
  RDW - Week 52 | 0.07 (0.141) | 0.35 (0.582)

49. Secondary Outcome: Laboratory Values - CMP (g/dL)
Description: Changes from baseline in CMP laboratory values with unit of g/dL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
g/dL
  Albumin - Baseline | 4.70 (0.089) | 4.64 (0.071)
  Albumin - Week 24: number analyzed (Participants) | 12 | 10
  Albumin - Week 24 | -0.03 (0.093) | -0.03 (0.122)
  Albumin - Week 52: number analyzed (Participants) | 11 | 10
  Albumin - Week 52 | 0.00 (0.086) | -0.03 (0.091)
  Calc Globulin - Baseline | 2.53 (0.100) | 2.10 (0.072)
  Calc Globulin - Week 24: number analyzed (Participants) | 12 | 10
  Calc Globulin - Week 24 | -0.14 (0.075) | -0.06 (0.072)
  Calc Globulin - Week 52: number analyzed (Participants) | 11 | 10
  Calc Globulin - Week 52 | -0.14 (0.059) | -0.05 (0.064)
  Protein - Baseline | 7.23 (0.120) | 6.74 (0.100)
  Protein - Week 24: number analyzed (Participants) | 12 | 10
  Protein - Week 24 | -0.17 (0.140) | -0.09 (0.146)
  Protein - Week 52: number analyzed (Participants) | 11 | 10
  Protein - Week 52 | -0.14 (0.106) | -0.08 (0.085)

50. Secondary Outcome: Laboratory Values - CMP (Ratio: Albumin (g/dL) to Calc. Globulin (g/dL))
Description: Changes from baseline in CMP laboratory values with units of Ratio: Albumin(g/dL) to Calc. Globulin(g/dL)
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: Ratio: Albumin(g/dL) to Globulin(g/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Ratio: Albumin(g/dL) to Globulin(g/dL
  Calc A/G - Baseline | 1.89 (0.086) | 2.23 (0.086)
  Calc A/G - Week 24: number analyzed (Participants) | 12 | 10
  Calc A/G - Week 24 | 0.10 (0.066) | 0.08 (0.100)
  Calc A/G - Week 52: number analyzed (Participants) | 11 | 10
  Calc A/G - Week 52 | 0.11 (0.076) | 0.04 (0.090)

51. Secondary Outcome: Laboratory Values - CMP (U/L)
Description: Changes from baseline in CMP laboratory values with units of U/L.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
U/L
  Alkaline Phosphatase - Baseline | 77.5 (9.35) | 69.0 (4.11)
  Alkaline Phosphatase - Week 24: number analyzed (Participants) | 12 | 10
  Alkaline Phosphatase - Week 24 | -2.6 (4.67) | -0.3 (2.48)
  Alkaline Phosphatase - Week 52: number analyzed (Participants) | 11 | 10
  Alkaline Phosphatase - Week 52 | 5.5 (4.75) | 1.0 (1.93)
  ALT - Baseline | 23.9 (2.66) | 17.7 (1.05)
  ALT - Week 24: number analyzed (Participants) | 12 | 10
  ALT - Week 24 | -1.4 (1.94) | 2.9 (1.97)
  ALT - Week 52: number analyzed (Participants) | 11 | 10
  ALT - Week 52 | 1.9 (4.03) | -0.1 (1.51)
  AST - Baseline | 25.7 (2.56) | 18.3 (1.50)
  AST - Week 24: number analyzed (Participants) | 12 | 10
  AST - Week 24 | -3.1 (2.07) | 2.1 (1.92)
  AST - Week 52: number analyzed (Participants) | 11 | 10
  AST - Week 52 | -2.8 (2.91) | -0.8 (1.10)

52. Secondary Outcome: Laboratory Values - CMP (mg/dL)
Description: Changes from baseline in CMP laboratory values with units of mg/dL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
mg/dL
  Bilirubin - Baseline | 0.41 (0.045) | 0.44 (0.051)
  Bilirubin - Week 24: number analyzed (Participants) | 12 | 10
  Bilirubin - Week 24 | 0.01 (0.060) | 0.15 (0.062)
  Bilirubin - Week 52: number analyzed (Participants) | 11 | 10
  Bilirubin - Week 52 | -0.02 (0.038) | 0.09 (0.062)
  Calcium - Baseline | 9.78 (0.099) | 9.51 (0.108)
  Calcium - Week 24: number analyzed (Participants) | 12 | 10
  Calcium - Week 24 | -0.20 (0.145) | -0.15 (0.134)
  Calcium - Week 52: number analyzed (Participants) | 11 | 10
  Calcium - Week 52 | -0.11 (0.110) | -0.03 (0.128)
  Creatinine - Baseline | 0.756 (0.0453) | 0.827 (0.0472)
  Creatinine - Week 24: number analyzed (Participants) | 12 | 10
  Creatinine - Week 24 | 0.008 (0.0288) | -0.000 (0.0278)
  Creatinine - Week 52: number analyzed (Participants) | 11 | 10
  Creatinine - Week 52 | -0.001 (0.0262) | 0.024 (0.0348)
  BUN - Baseline | 14.3 (1.31) | 13.4 (1.20)
  BUN - Week 24: number analyzed (Participants) | 12 | 10
  BUN - Week 24 | -0.5 (1.05) | 0.6 (1.25)
  BUN - Week 52: number analyzed (Participants) | 11 | 10
  BUN - Week 52 | 1.5 (0.86) | -0.1 (1.09)
  Glucose - Baseline | 95.3 (3.58) | 94.1 (2.04)
  Glucose - Week 24: number analyzed (Participants) | 12 | 10
  Glucose - Week 24 | -1.9 (3.45) | -3.6 (3.77)
  Glucose - Week 52: number analyzed (Participants) | 11 | 10
  Glucose - Week 52 | 2.5 (1.83) | -1.6 (3.81)

53. Secondary Outcome: Laboratory Values - CMP (mEq/L)
Description: Changes from baseline in CMP laboratory values with units of mEq/L.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
mEq/L
  Chloride - Baseline | 103.5 (0.97) | 103.7 (0.81)
  Chloride - Week 24: number analyzed (Participants) | 12 | 10
  Chloride - Week 24 | -0.3 (0.71) | 1.4 (0.83)
  Chloride - Week 52: number analyzed (Participants) | 11 | 10
  Chloride - Week 52 | 0.2 (0.64) | 0.8 (1.10)
  Carbon Dioxide - Baseline | 25.2 (0.76) | 24.7 (0.63)
  Carbon Dioxide - Week 24: number analyzed (Participants) | 12 | 10
  Carbon Dioxide - Week 24 | 0.1 (0.58) | 0.1 (0.72)
  Carbon Dioxide - Week 52: number analyzed (Participants) | 11 | 10
  Carbon Dioxide - Week 52 | 0.5 (0.39) | 0.1 (0.86)
  Potassium - Baseline | 4.47 (0.128) | 4.31 (0.061)
  Potassium - Week 24: number analyzed (Participants) | 12 | 10
  Potassium - Week 24 | -0.22 (0.135) | -0.13 (0.060)
  Potassium - Week 52: number analyzed (Participants) | 11 | 10
  Potassium - Week 52 | -0.11 (0.164) | -0.11 (0.077)
  Sodium - Baseline | 142.0 (0.76) | 140.5 (0.53)
  Sodium - Week 24: number analyzed (Participants) | 12 | 10
  Sodium - Week 24 | -0.9 (0.85) | 1.0 (0.47)
  Sodium - Week 52: number analyzed (Participants) | 11 | 10
  Sodium - Week 52 | -0.4 (0.51) | 0.7 (0.82)

54. Secondary Outcome: Laboratory Values - CMP (mL/Min/1.73m^2)
Description: Changes from baseline in CMP laboratory values with units of mL/min/1.73m^2.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
mL/min/1.73m^2
  Glomerular Filtration Rate (eGFR) - Baseline | 99.5 (2.41) | 94.4 (5.65)
  Glomerular Filtration Rate (eGFR) - Week 24: number analyzed (Participants) | 12 | 10
  Glomerular Filtration Rate (eGFR) - Week 24 | -1.7 (2.28) | 0.2 (3.18)
  Glomerular Filtration Rate (eGFR) - Week 52: number analyzed (Participants) | 11 | 10
  Glomerular Filtration Rate (eGFR) - Week 52 | -0.8 (1.75) | -2.7 (3.99)

55. Secondary Outcome: Laboratory Values - CMP (Ratio: Urea Nitrogen (mg/dL) to Creatinine (mg/dL))
Description: Changes from baseline in CMP laboratory values with units of Ratio: Urea Nitrogen (mg/dL) to Creatinine (mg/dL).
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: Ratio:Urea nit.(mg/dL) /creatinin(mg/dL)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Ratio:Urea nit.(mg/dL) /creatinin(mg/dL)
  Calc BUN/Creat - Baseline | 19.7 (2.44) | 16.3 (1.00)
  Calc BUN/Creat - Week 24: number analyzed (Participants) | 12 | 10
  Calc BUN/Creat - Week 24 | -0.6 (1.43) | 0.4 (1.61)
  Calc BUN/Creat - Week 52: number analyzed (Participants) | 11 | 10
  Calc BUN/Creat - Week 52 | 2.5 (1.15) | -0.6 (1.59)

56. Secondary Outcome: Laboratory Values - Coagulation Panel (Seconds)
Description: Changes from baseline in Coagulation Panel values with units of seconds.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Seconds
  Prothrombin Time (PT) - Baseline | 12.95 (0.183) | 13.23 (0.152)
  Prothrombin Time (PT) - Week 24: number analyzed (Participants) | 12 | 10
  Prothrombin Time (PT) - Week 24 | 1.00 (0.833) | 0.08 (0.096)
  Prothrombin Time (PT) - Week 52: number analyzed (Participants) | 11 | 10
  Prothrombin Time (PT) - Week 52 | 1.28 (1.064) | 0.12 (0.049)
  PTT - Baseline | 29.78 (1.056) | 30.06 (0.618)
  PTT - Week 24: number analyzed (Participants) | 12 | 10
  PTT - Week 24 | 0.73 (0.936) | -0.88 (0.528)
  PTT - Week 52: number analyzed (Participants) | 11 | 10
  PTT - Week 52 | 2.63 (1.712) | -1.22 (0.707)

57. Secondary Outcome: Laboratory Values. Coagulation Panel (Ratio: Prothrombin Time (Seconds) / Mean Normal Prothrombin Time (Seconds))
Description: Changes from baseline in Coagulation laboratory values with units of Ratio: Prothrombin time (seconds) / Mean normal prothrombin time (seconds).
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: Ratio: PT (seconds) / MNPT (seconds)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 12
Ratio: PT (seconds) / MNPT (seconds)
  INR - Baseline | 0.94 (0.019) | 0.96 (0.015)
  INR - Week 24: number analyzed (Participants) | 12 | 10
  INR - Week 24 | 0.11 (0.092) | 0.04 (0.016)
  INR - Week 52: number analyzed (Participants) | 11 | 10
  INR - Week 52 | 0.14 (0.119) | 0.02 (0.013)

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) through End of Study (Week 52)
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12) | Placebo (N=12)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Cellulitis of arm (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12) | Placebo (N=12)
Headache (Nervous system disorders) | 8 (16) | 5 (15)
Muscle spasticity (Nervous system disorders) | 0 (0) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Multiple Sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (5)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
White matter lesion (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 5 (10)
Feeling abnormal (General disorders) | 1 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 1 (2) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Muscle strength abnormal (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT05116540/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT05116540/SAP_001.pdf